CLINICAL TRIAL: NCT04183634
Title: An Open, Randomised, Single Dose, 2-period, 2-sequence Crossover Adhesion Study of Two Different Transdermal Patches Containing Rotigotine.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-06-TTS-10
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
Keywords: adhesiveness
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: Rotigotine TTS (Test) - Period 2: Neupro (Reference) (Experimental): For each period: an 18 mg transdermal patch to deliver 8 mg/24h will be applied for 24 h
  Interventions: Drug: Rotigotine TTS (Test); Drug: Neupro (Reference)
- Period 1: Neupro (Reference) - Period 2: Rotigotine TTS (Test) (Active Comparator): For each period: an 18 mg transdermal patch to deliver 8 mg/24h will be applied for 24 h
  Interventions: Drug: Rotigotine TTS (Test); Drug: Neupro (Reference)

INTERVENTIONS:
Drug: Rotigotine TTS (Test) — Transdermal patch containing Rotigotine 18 mg to deliver 8 mg/24.
Drug: Neupro (Reference) — Neupro®: transdermal patch containing Rotigotine 18 mg to deliver 8 mg/24 h.

SUMMARY:
The objective of this study is to evaluate the adhesion of the test product when compared to the reference product following a single transdermal application.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the adhesion of the test product when compared to the reference product following a single transdermal application.

The following evaluations will be assessed as "yes" or "no":

* Cold flow (dark ring formed around the patch)
* Patch movement/displacement
* Patch wrinkling
* Residue formation (at patch application on the release liner and at patch removal on the skin) Safety and tolerability of a single dose application of a patch containing 18 mg rotigotine (Test) against a patch containing 18 mg rotigotine (Reference) will be evaluated in terms of vital signs and AEs.

AEs and clinical tolerability will be monitored at all clinical trial visits. The safety evaluation will be based upon the review of the individual values (potentially clinically important abnormalities) and descriptive statistics (summary tables, graphics).

As additional safety parameters for the clinical trial physical examination findings, clinical laboratory parameters, and 12-lead ECGs will be assessed at the screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic Parkinson's Disease assessed as eligible for receiving 18 mg/IRR 8 mg/24 h rotigotine via the test and the reference product each on subsequent days in order to reach the dose of active substance at the individual routine medical care. Patients should be on a stable rotigotine dose of at least 8 mg/24 h for at least 1 week before screening.

Exclusion Criteria:

* Current participation in another clinical trial, participation in another clinical study (i.e. last protocol specified visit) involving another IMP within at least 28 days prior to first application or previous participation in this clinical Trial
* History or presence of clinically significant dermatologic diseases or conditions, such as atopy, neurodermatitis, contact allergy, eczema, psoriasis, vitiligo, melanoma, squamous cell carcinoma.
* History or presence of any dermatological condition or skin sensitivity that could affect IMP Absorption
* History of clinically relevant (severe) hypersensitivity to the active pharmaceutical ingredient or substances of the same class or one of the excipients, clinically relevant allergy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Patch Adhesion | 24 hours in each Treatment Period
  Patch Adhesion will be measured as the percentage of area that remained adhered after 24 hours of patch application.

SECONDARY OUTCOMES:
Number of patients with cold flow | 24 hours in each Treatment Period
  Cold flow is defined as dark ring formed around the patch
Number of patients with patch movement/displacement | 24 hours in each Treatment Period
Number of patients with patch wrinkling | 24 hours in each Treatment Period
Number of patients with patch residue formation | 24 hours in each Treatment Period
  Patch residue formation is assessed at patch application on the release liner and at patch removal on the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (1):
- Sandoz Investigative Site, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No